CLINICAL TRIAL: NCT04733612
Title: Effects of Short-Message Notifications on Medication Adherence, Physical Activity and Fasting Blood Glucose Control and Correlation of These With the Health-Related Quality of Life in Mid-aged Diabetic Patients
Brief Title: The Effects of Short Message Notifications on Middle-Aged Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Bernard Tahirbegolli, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20135
Record Dates: First submitted 2021-01-16; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Type2 Diabetes Mellitus
Keywords: Diabetes mellitus; Public health
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS Group (Experimental): In addition to traditional treatment received three to four informative SMS messages per week during the 6-month period
  Interventions: Other: Informative messages
- Control Group (No Intervention): Followed in accordance with the traditional treatment schedule

INTERVENTIONS:
Other: Informative messages — In addition to their standard treatments, an informative SMS (text message) on diabetes was sent to the intervention group three to four times a week for six months.
  The short messages were in the form of a short sentence for the subject and the predicate. The messages sent have been prepared in such a way that they do not exceed 1 SMS quota and are less than 160 characters on mobile phones.
  Arms: SMS Group

SUMMARY:
The objective of our study was to assess awareness-raising of medication adherence (MA), physical activity (PA), fasting blood glucose (FBG), and glycated hemoglobin A (HbA1c) values by providing information on diabetes via short message (SMS) technology.

DETAILED DESCRIPTION:
The study investigates T2DM patients who have not had surgery or cardiac event in the last 3 months, between the ages of 40 and 64 years, with T2DM diagnosis between the last 1 and 10 years and oral antidiabetic therapy for at least 1 The study design is a single-blinded randomized, controlled study, and was conducted in the Diabetes Polyclinic of the Istanbul University Medical Faculty Hospital.

Patients randomly assigned to the intervention group, in addition to traditional treatment received three to four informative SMS messages per week during the 6-month period, while the control group was followed in accordance with the traditional treatment schedule.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 Diabetes Mellitus (T2DM) between the last 1 and 10 years
* Being aged between 40 and 64 years old,
* Is treated for a minimum of 1 year with at least one oral antidiabetic drug.

Exclusion Criteria:

* Clinical diagnosis of T2DM for less than 1 year or more than 10 years.
* Those who have had surgery or a cardiac event in the last 3 months or during the investigation.
* Those under 40 and over 64 years of age.
* Patients with T2DM that have not been treated with oral antidiabetic medication.
* Volunteers who once did not participate in the control examinations in both groups were excluded from the evaluation.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-02-26 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose | Beginning
  After 8 hours of fasting in the morning, venous whole blood samples were taken to yellow capped tubes for fasting blood glucose (mmol/dL).
Change from Baseline Fasting blood glucose at 3 months | 3 months after beginning
  After 8 hours of fasting in the morning, venous whole blood samples were taken to yellow capped tubes for fasting blood glucose (mmol/dL).
Change from Baseline Fasting blood glucose at 6 months | 6 months after beginning
  After 8 hours of fasting in the morning, venous whole blood samples were taken to yellow capped tubes for fasting blood glucose (mmol/dL).
Glycated hemoglobin A (HbA1c) | Beginning
  In the HbA1c evaluation (%), after 8 hours of fasting by volunteers, venous whole blood samples were taken in purple tubes (EDTA) between 08:00 and 10:00 a.m. and evaluated by the HPLC method.
Change from Baseline of Glycated hemoglobin A (HbA1c) at 3 months | 3 months after beginning
  In the HbA1c evaluation (%), after 8 hours of fasting by volunteers, venous whole blood samples were taken in purple tubes (EDTA) between 08:00 and 10:00 a.m. and evaluated by the HPLC method
Change from Baseline of Glycated hemoglobin A (HbA1c) at 6 months | 6 months after beginning
  In the HbA1c evaluation (%), after 8 hours of fasting by volunteers, venous whole blood samples were taken in purple tubes (EDTA) between 08:00 and 10:00 a.m. and evaluated by the HPLC method
Physical Activity level | Beginning
  The International Physical Activity Questionnaire (IPAQ) was used to evaluate the physical activity level of the participants at the beginning of the study.
  This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting. The higher scores mean a better outcome.
Change from Baseline Physical Activity at 3 months | 3 months from beginning
  The International Physical Activity Questionnaire (IPAQ) was used to evaluate the physical activity level of the participants at at 3 months after the beginning of the study.
  This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting. The higher scores mean a better outcome.
Change from Baseline Physical Activity at 6 months | 6 months from beginning
  The International Physical Activity Questionnaire (IPAQ) was used to evaluate the change in physical activity level of the participants at at 6 months after the beginning of the study.
  This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting. The higher scores mean a better outcome.
Drug Adherence | Beginning
  The Morisky Medication Adherence Scale (MMAS-8) was used to assess the compliance of patients with drug treatment.
  If the patient scores higher on the scale, they will be assessed as more adherent. If they score lower on the scale, they are presumed to be struggling with non-adherence.
Change from Baseline Drug Adherence at 3 months | 3 months after beginning
  The Morisky Medication Adherence Scale was used to assess the compliance of patients with drug treatment.
  If the patient scores higher on the scale, they will be assessed as more adherent. If they score lower on the scale, they are presumed to be struggling with non-adherence.
Change from Baseline Drug Adherence at 6 months | 6 months after beginning
  The Morisky Medication Adherence Scale (MMAS-8) was used to assess the compliance of patients with drug treatment.
  If the patient scores higher on the scale, they will be assessed as more adherent. If they score lower on the scale, they are presumed to be struggling with non-adherence.
Quality of Life Assessed by SF-36v2 | Beginning
  The Short-Form Health Survey (SF-36v2) is used to asses the quality of life of volunteers'. It has 36 items grouped in 8 dimensions: physical functioning, physical and emotional limitations, social functioning, bodily pain, general and mental health. The higher scores mean a better outcome.
Change from Baseline Quality of Life Assessed by SF-36v2 at 3 months | 3 months after beginning
  The Short-Form Health Survey (SF-36v2) is used to asses the quality of life of volunteers'. It has 36 items grouped in 8 dimensions: physical functioning, physical and emotional limitations, social functioning, bodily pain, general and mental health. The higher scores mean a better outcome.
Change from Baseline Quality of Life Assessed by SF-36v2 at 6 months | 6 months after beginning
  The Short-Form Health Survey (SF-36v2) is used to asses the quality of life of volunteers'. It has 36 items grouped in 8 dimensions: physical functioning, physical and emotional limitations, social functioning, bodily pain, general and mental health. The higher scores mean a better outcome.

SECONDARY OUTCOMES:
Baseline blood pressure | Beginning
  The volunteers' systolic and diastolic blood pressure (mmHg) was measured by a physician through a manual cuff and stethoscope after sitting for at least 5 minutes, from the left arm at the level of the heart, as suggested in the literature.
Change from Baseline blood pressure at 3 months | 3 months after beginning
  The volunteers' systolic and diastolic blood pressure (mmHg) was measured by a physician through a manual cuff and stethoscope after sitting for at least 5 minutes, from the left arm at the level of the heart, as suggested in the literature.
Change from Baseline blood pressure at 6 months | 6 months after beginning
  The volunteers' systolic and diastolic blood pressure (mmHg) was measured by a physician through a manual cuff and stethoscope after sitting for at least 5 minutes, from the left arm at the level of the heart, as suggested in the literature.
Baseline heart rate | Beginning
  The volunteers' heart rate count was measured by a finger-type pulse oximeter, from the index finger of the right or left hand after resting for at least 5 minutes.
Change from Baseline heart rate at 3 months | 3 Months After Beginning
  The volunteers' heart rate count was measured by a finger-type pulse oximeter, from the index finger of the right or left hand after resting for at least 5 minutes.
Change from Baseline heart rate at 6 months | 6 Months After Beginning
  The volunteers' heart rate count was measured by a finger-type pulse oximeter, from the index finger of the right or left hand after resting for at least 5 minutes.
Baseline Body Mass Index | Beginning
  The height (cm) of the volunteers was obtained in the morning, after 8 hours of fasting, without shoes, standing upright, by measuring the distance from the top of the head to the floor with a calibrated stadiometer. Body weight (kg) were measured in the morning after 8 hours of fasting, with light clothing and bare feet, with a calibrated and valid 'Tanita Body Composition Analyzer TBF-410GS' brand bioelectrical impedance analyzer.
  Body Mass Index (BMI) is calculated using a person's height and weight as shown in formula:
  BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in meter square.
Change from Baseline Body Mass Index at 3 months | 3 months after Beginning
  The height (cm) of the volunteers was obtained in the morning, after 8 hours of fasting, without shoes, standing upright, by measuring the distance from the top of the head to the floor with a calibrated stadiometer. Body weight (kg) were measured in the morning after 8 hours of fasting, with light clothing and bare feet, with a calibrated and valid 'Tanita Body Composition Analyzer TBF-410GS' brand bioelectrical impedance analyzer.
  Body Mass Index (BMI) is calculated using a person's height and weight as shown in formula:
  BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in meter square.
Change from Baseline Body Mass Index at 6 months | 6 months after Beginning
  The height (cm) of the volunteers was obtained in the morning, after 8 hours of fasting, without shoes, standing upright, by measuring the distance from the top of the head to the floor with a calibrated stadiometer. Body weight (kg) were measured in the morning after 8 hours of fasting, with light clothing and bare feet, with a calibrated and valid 'Tanita Body Composition Analyzer TBF-410GS' brand bioelectrical impedance analyzer.
  Body Mass Index (BMI) is calculated using a person's height and weight as shown in formula:
  BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in meter square.
Baseline body fat ratios | Beginning
  The body fat ratios were measured in the morning after 8 hours of fasting, with light clothing and bare feet, with a calibrated and valid 'Tanita Body Composition Analyzer TBF-410GS' brand bioelectrical impedance analyzer.
Change from Baseline Body Fat Ratios at 3 Months | 3 Months After Beginning
  The body fat ratios were measured in the morning after 8 hours of fasting, with light clothing and bare feet, with a calibrated and valid 'Tanita Body Composition Analyzer TBF-410GS' brand bioelectrical impedance analyzer.
Change from Baseline Body Fat Ratios at 6 Months | 6 Months After Beginning
  The body fat ratios were measured in the morning after 8 hours of fasting, with light clothing and bare feet, with a calibrated and valid 'Tanita Body Composition Analyzer TBF-410GS' brand bioelectrical impedance analyzer.
Baseline waist/hip ratio | Beginning
  The volunteers waist and hip circumference and waist/hip ratio were measured by tape measure after 8 hours of fasting in the morning with thin clothes on them.
  Waist circumference (cm) was measured at the level of the umbilicus and hip circumference (cm) at the level of the femur trochanter major.
  Waist/hip ratio (WHR) were were calculated as follows
  waist/hip ratio= waist circumference / hip circumference
Change from Baseline waist/hip ratio at 3 Months | 3 Months after Beginning
  The volunteers waist and hip circumference and waist/hip ratio were measured by tape measure after 8 hours of fasting in the morning with thin clothes on them.
  Waist circumference (cm) was measured at the level of the umbilicus and hip circumference (cm) at the level of the femur trochanter major.
  Waist/hip ratio (WHR) were were calculated as follows
  waist/hip ratio= waist circumference / hip circumference
Baseline Diet and Nutritional Habits | Beginning
  The last three days' food intake form is used to collect the information about daily nutritional habits of volunteers'. The amount of food and the frequency are marked.
Change from Baseline Diet and Nutritional Habits at 3 months | 3 Months after Beginning
  The last three days' food intake form is used to collect the information about daily nutritional habits of volunteers'. The amount of food and the frequency are marked.
Change from Baseline Diet and Nutritional Habits at 6 months | 6 Months after Beginning
  The last three days' food intake form is used to collect the information about daily nutritional habits of volunteers'. The amount of food and the frequency are marked.
Baseline Energy Intake | Beginning
  From the last three days' food intake form the average calories (kcal) of macro and micronutrients are calculated.
Change from Baseline Energy Intake at 3 months | 3 months after Beginning
  From the last three days' food intake form the average calories (kcal) of macro and micronutrients are calculated.
Change from Baseline Energy Intake at 6 months | 6 months after Beginning
  From the last three days' food intake form the average calories (kcal) of macro and micronutrients are calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Suphi Vehid, Prof. Dr., Study Chair — Istanbul University

IPD SHARING:
Plan to Share IPD: No
Since the start date of the study is before 18 January 2017, individual participant data (IPD) will only be available to other researchers on a reasonable request.

REFERENCES:
- [Derived] Tahirbegolli B, Tahirbegolli IA, Cakmak R, Idiz C, Cavdar S, Bagdemir E, Vehid S. Effects of Short-message Notifications on Type 2 Diabetes Management in Middle-aged Turkish Patients: A Randomized Trial. Balkan Med J. 2022 Mar 14;39(2):161-162. doi: 10.4274/balkanmedj.galenos.2021.2021-10-47. No abstract available. PMID 35330570